CLINICAL TRIAL: NCT03018678
Title: Screening Protocol for a Gene Therapy Trial in Subjects With Homozygous Familial Hypercholesterolemia
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 822899
Record Dates: First submitted 2017-01-10; First posted 2017-01-12 (Estimated); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Hypercholesterolemia, Familial
MeSH Terms: conditions — Hyperlipoproteinemia Type II

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Nab titer samples are retained, but there is no potential for DNA extraction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with HOFH: No intervention

SUMMARY:
The purpose of this protocol is to identify and screen potential candidates for future enrollment in a gene therapy clinical trial for HoFH.

DETAILED DESCRIPTION:
Homozygous Familial Hypercholesterolemia (HoFH) is a rare genetic metabolic disorder characterized by markedly elevated LDL-cholesterol (LDL-C) levels, resulting in severe atherosclerosis often leading to early onset of cardiovascular disease. The most frequent cause is mutation in the LDL receptor gene (LDLR). LDL-C levels remain frequently above acceptable levels despite treatment with multiple existing lipid lowering drugs and/or LDL apheresis. Thus, the functional replacement of the defective LDLR via AAV-based liver-directed gene therapy may be a viable approach to treat this disease and improve response to current lipid-lowering treatments. The purpose of this protocol is to identify and screen potential candidates for future enrollment in a gene therapy clinical trial. No study drug will be administered in this screening study.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 years of age
* Clinical presentation consistent with homozygous FH
* Subjects must be able to comprehend and willing to provide a signed IRB approved Informed Consent Form

Exclusion Criteria:

* Known to carry confirmed mutations in genes affecting LDL receptor functionality other than the LDLR gene
* History of cirrhosis based on documented histological evaluation or non-invasive imaging
* Documented diagnosis of any of the following liver diseases: Hepatitis B or C; Biopsy-proven nonalcoholic steatohepatitis; Biopsy-proven alcoholic liver disease; Autoimmune hepatitis; Primary biliary cirrhosis; Primary sclerosing cholangitis; Wilson's disease; Hemochromatosis; alpha1 anti-trypsin deficiency
* History of immunodeficiency diseases, including a positive HIV test result
* Previous organ transplantation
* Serious or unstable medical or psychological conditions that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study
* Inability to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinical diagnosis compatible with homozygous familial hypercholesterolemia (HoFH)
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2016-03; Primary Completion 2017-05-30 (Actual); Study Completion 2019-12-03 (Actual)

PRIMARY OUTCOMES:
genetic analysis | Screening phase
  identification of genetic, confirmation of FH
Neutralizing antibodies | Screening phase
  identification of subjects with no or minimal neutralizing antibodies titer <= 1:10

CONTACTS AND LOCATIONS:
Overall Officials: Marina Cuchel, MD, PhD, Principal Investigator — Associate Professor
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The following entities may use or share information: (1) the investigator for the study and the study team, (2) the University of Pennsylvania Institutional Review Boards (the committees who oversee research on human subjects) and University of Pennsylvania Office of Regulatory Affairs, (3) The University of Pennsylvania Office of Clinical Research (the office which monitors research studies), and (4) authorized members of the University of Pennsylvania and the University of Pennsylvania Health System and School of Medicine workforce who may need to access your information in the performance of their duties (for example: to provide treatment, to ensure integrity of the research, accounting or billing matters, etc).
Time Frame: Has been open until 2015. Data is open until decided.
Access Criteria: Data will be de-identified prior to sharing with other entities.